CLINICAL TRIAL: NCT04687241
Title: Efficacy and Safety of Almonertinib Versus Placebo as Adjuvant Therapy for Subjects With Resected Stage II-IIIB NSCLC Harboring EGFR-sensitive Mutations: A Randomized, Controlled, Double-blind, Phase 3 and Multicenter Clinical Study
Brief Title: Almonertinib Versus Placebo as Adjuvant Therapy in Resected Stage II-IIIB Non-Small Cell Lung Cancer With EGFR-sensitive Mutations
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-10296-302
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib (Experimental)
  Interventions: Drug: Almonertinib
- Placebo Almonertinib (Placebo Comparator)
  Interventions: Drug: Placebo Almonertinib

INTERVENTIONS:
Drug: Almonertinib — The initial dose of Almonertinib 110 mg daily can be reduced to 55 mg daily under specific conditions.
  Other Names: HS-10296
  Arms: Almonertinib
Drug: Placebo Almonertinib — Placebo Almonertinib
  Arms: Placebo Almonertinib

SUMMARY:
To assess the efficacy and safety of Almonertinib versus placebo in patients with epidermal growth factor receptor mutation-positive (EGFRm+) stage II-IIIB non-small cell lung cancer (NSCLC), following complete tumor resection with or without adjuvant chemotherapy.

DETAILED DESCRIPTION:
HS-10296-302 is a randomized, placebo-controlled, double-blind, multicenter, phase III study to assess the efficacy and safety of Almonertinib versus placebo in stage II-IIIB NSCLC with EGFRm+ following complete tumor resection, with or without postoperative adjuvant chemotherapy (2~4 cycles of platinum-based doublet). Eligible patients are randomized to receive either Almonertinib (110 mg orally, once daily) or placebo (110 mg orally, once daily) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of informed consent before any study-specific procedures, sampling and analyses.

  2. Male or female, age at least 18 years. 3. Histologically confirmed diagnosis of primary non-small lung cancer (NSCLC) on predominantly non-squamous histology.

  4. MRI or CT scan of the brain must be done before surgery to exclude brain metastasis.

  5. Complete surgical resection of the primary NSCLC and lymphadenectomy are mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumor.

  6. Patients must be classified post-operatively as Stage IIA, IIB, IIIA or IIIB (only T3N2M0) based on pathologic criteria.

  7. Confirmation by the central laboratory that the tumor harbors one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations including T790M.

  8. Complete recovery from surgery and standard post-operative therapy (if applicable) at the time of randomization.

  9. A WHO performance status of 0-1 with no deterioration over the past 2 weeks and a minimum life expectancy of 12 weeks.

  10. Female patients should be using adequate contraceptive measures and should not be breastfeeding at the screening period, during the study, and six months after the last dosing of study. A pregnancy test should be done before first dosing unless having evidence of non-child-bearing potential.

  11. Male patients should be willing to use barrier contraception (condoms).

Exclusion Criteria:

* 1. Patients who have had only segmentectomies or wedge resections. 2. Treatment with any of the following:

  1. Any prior anticancer therapy for the current lung cancer (pre-operative (neoadjuvant) platinum-based or other chemotherapy, pre-operative or post-operative or planned radiation therapy, neoadjuvant or adjuvant EGFR-TKI, other targeted therapy and immunotherapy).
  2. Major surgery (including primary tumor surgery, excluding placement of vascular access) within 3 weeks of the first dose of study drug.
  3. Patients currently receiving medications or herbal supplements known to be strong inducers and inhibitors of cytochrome P450 (CYP) 3A4.
  4. Treatment with an investigational drug within five half-lives of the compound or any of its related material.

     3. Inadequate bone marrow reserve or organ function. 4. Any of the following cardiac criteria:

  <!-- -->

  1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., PR interval > 250 ms).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure or any concomitant medication known to prolong the QT interval.
  4. Left ventricular ejection fraction (LVEF) ≤ 40%. 5. History of other malignancies, excluding full treated non-melanoma skin cancer, in-situ cancer, or other solid tumors that hadn't recurrent for > 5 years following the end of treatment.

     6. Any evidence of severe or uncontrolled systemic diseases (including uncontrolled hypertension and active bleeding diatheses) or active infection (including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV)).

     7. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow the study drug that would preclude adequate absorption of Almonertinib.

     8. History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.

     9. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 except alopecia and Grade 2 prior platinum-therapy related neuropathy.

     10. History of hypersensitivity to any active or inactive ingredient of Almonertinib or to drugs with a similar chemical structure or class to Almonertinib.

     11. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply study procedures, restrictions, and requirements.

     12. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.

     13. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
DFS (Disease free survival) assessed by IRC (Independent Review Committee) | From the time of randomization to recurrence of tumor or death, approximately 4 years.
  DFS is defined as the time from randomization to the recurrence of tumor as assessed by IRC or death from any cause on study. The patients will receive long-term follow-up including chest and abdominal CT every 12 weeks during Year 1, then every 24 weeks during Years 2 to 5, and every 48 weeks during Year 6 and onwards; MRI/CT of brain, and bone scan performed every 48 weeks.

SECONDARY OUTCOMES:
DFS (Disease free survival) assessed by INVs (Investigators) | From the time of randomization to recurrence of tumor or death, approximately 4 years.
  The patients will receive long-term follow-up including chest and abdominal CT every 12 weeks during Year 1, then every 24 weeks during Years 2 to 5, and every 48 weeks during Year 6 and onwards; MRI/CT of brain, and bone scan performed every 48 weeks. DFS is defined as the time from randomization to the recurrence of tumor as assessed by INVs or death from any cause on study.
DFS rate at 2, 3 and 5 years assessed by IRC | From the time of randomization to recurrence of tumor or death, approximately 6 years.
  Defined as the proportion of patients alive and disease free at 2, 3 and 5 years, respectively, estimated from Kaplan Meier plots of the primary endpoint of DFS at the time of the primary analysis.
OS (Overall survival) | The time from randomization to death due to any cause, approximately 8 years.
  OS is deﬁned as the time from randomization to death due to any cause. The survival will be followed up with telephone every 24 weeks after discontinuation of the randomized treatment.
OS rate at 5 years | The time from randomization to death due to any cause, approximately 8 years.
  OS rate at 5 years is defined as the proportion of patients alive at 5 years.
Incidence and severity of adverse events (AEs) | From the screening period to 28 days after treatment completion, approximately 4 years.
  AEs are graded according to CTCAE v5.0 and recorded in the case report form.
Plasma concentrations of Almonertinib and HAS-719 metabolite. | From Cycle 3 (Each cycle =3 weeks) to Cycle 4, approximately 3 weeks.
  Defined as the pharmacokinetics exposure parameters derived from plasma concentrations of Almonertinib and its metabolite, HAS-719.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, MD, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Province Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang L, Zhang X, Wu L, Xing W, Liu C, Zhang P, Chen K, Shi J, Xu S, Zhang X, Dong X, Fang H, Yu X, Gao Y, Li G, Chen Z, Fan S, Zhang X, Cheng Y. Aumolertinib as adjuvant therapy in resected EGFR-mutated non-small-cell lung cancer (ARTS): a double-blind, multicentre, randomised, controlled, phase 3 trial. Lancet Oncol. 2026 Jan 12:S1470-2045(25)00643-6. doi: 10.1016/S1470-2045(25)00643-6. Online ahead of print. PMID 41539318